CLINICAL TRIAL: NCT05574023
Title: Impact of Continuous Glucose Monitoring (CGM) With Predictive Alarm for Hypoglycemia (Guardian Connect System) on Glycemic Control and Hypoglycemia Management in a Group of Adolescents With Type 1 Diabetes Mellitus Treated With Multiple Daily Insulin Injections (MDI).
Brief Title: Effect of CGM With Predictive Alarm on Hypoglycemia in Young Patients With T1D.
Acronym: CGMHYPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3142CESC
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a crossover, monocentric and randomized study with a post-market medical device.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predictive Alarm (PA) (Experimental): Patients use the CGM sensor with Predictive Alarm on set at 70 mg/dl in 20 minutes for hypoglycemia and at 250 mg/dl in 20 minutes for hyperglycemia.
  Interventions: Device: Use of Predictive Alarm for hypoglycaemia or hyperglycaemia
- Alarm on Threshold (AoT) (Active Comparator): Patients use the CGM sensor with alarms on a threshold of 70 mg/dl for hypoglycemia and 250 mg/dl for hyperglycemia.
  Interventions: Device: Use of Alarm on Threshold for hypoglycaemia or hyperglycaemia

INTERVENTIONS:
Device: Use of Predictive Alarm for hypoglycaemia or hyperglycaemia — Patients use CGM sensor with Predictive Alarm set at 70 mg/dl in 20 minutes for hypoglycemia and at 250 mg/dl in 20 minutes for hyperglycemia.
  1. in case of alarm from the hypoglycemia predictive algorithm, the indicated treatment was 0.1g of sugar/kg of body weight;
  2. in case of alarm from the hyperglycemia predictive algorithm, the indication was to give an extra shot of rapid-acting insulin. The dose will be calculated on the basis of personal insulin sensitivity factor (ISF), considering as target a blood glucose of 120 mg/dl and 250 mg/dl as the projected blood glucose level that will be reached in 20 minutes. This could be done only if there is no active insulin on-board, after at least 3 hours from the last rapid-acting insulin injection.
  Arms: Predictive Alarm (PA)
Device: Use of Alarm on Threshold for hypoglycaemia or hyperglycaemia — in case of alarm of hypoglycemia, the indicated treatment was 0.3g of sugar/kg of body weight, max 15g.
  in case of alarm of hyperglycemia, the indication will be to give an extra shot of rapid-acting insulin. The dose will be calculated on the basis of personal insulin sensitivity factor (ISF), considering as target a blood glucose of 120 mg/dl and 250 mg/dl as blood glucose level to correct. This could be done only if there is no active insulin on-board, after at least 3 hours from the last rapid-acting insulin injection.
  Arms: Alarm on Threshold (AoT)

SUMMARY:
The use of continuous glucose monitoring (CGM) is becoming the new standard in glycometabolic control in patients with Type 1 Diabetes Mellitus (T1DM) even in subjects in multiple daily insulin injections (MDI). Compared to self-monitoring of blood glucose (SMBG), the CGM systems allow continuous monitoring of the glycemic trends contributing to modify the therapeutic habits of adult and pediatric patients with T1DM and allowing to better managing of critical situations such as hypoglycemia. Recently, the accuracy and reliability performance of the latest generation of CGMs using predictive alarm for hypoglycaemia and hyperglycemia has been compared to other commercially available CGM systems, showing good levels of concordance.

The use of this new technology, through the continuous monitoring of the pre-and post-prandial glucose levels and the evaluation of the glycemic trends, could influence the therapeutic habits of patients and could substantially contribute to modifying insulin therapy. Furthermore, the presence of the predictive alarm technology for hypoglycemia could lead to reduce the number of hypoglycemic episodes and to modify the way these hypoglycemic episodes are managed; moreover, the use of this technology could improve the time spent in the target glycemic range [Time in Range (TIR), 70-180 mg/dl] with possible improvement also in glycemic variability control.

ELIGIBILITY:
Inclusion Criteria:

* T1DM for at least 12 months [assessed by positivity of at least one of the antibodies against islet cells (ICA), insulin (IAA), glutamate dehydroxylase (GADA), islet antigen 2 (IA2A), or Zinc Transporter 8 Antibodies (ZnT8)];
* MDI therapy from at least 6 months with basal-bolus treatment (long acting insulin analog plus rapid acting insulin analogue);
* HbA1c < 9.0%
* normal weight (BMI <85th percentile for age and gender);
* no other chronic diseases (thyroiditis, celiac disease, etc) or eating behavior disorders (DCA);
* signed informed consent from parents or legal guardians and patients (<18 y).

Exclusion Criteria:

* T1DM for less than 12 months;
* CSII therapy
* Previous usage of CGM with predictive alarm for hypoglycemia or hyperglycemia
* MDI therapy from less than 6 months
* use of regular insulin instead of rapid acting insulin analogue;
* other chronic diseases (thyroiditis, celiac disease, etc.) or eating behavior disorders (DCA).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Less time spent in hypoglycaemia using Predictive Alarm vs Alarm on Threshold | 2 weeks CGM data with PA vs 2 weeks CGM data with AoT
  the difference in the percentage of time spent below 70 mg/dl (TBR < 70 mg/dl) between the Alarm on Threshold (AoT) and the Predictive Alarm (PA) arms after 2 weeks of treatment

SECONDARY OUTCOMES:
Better glycemic metrics using Predictive Alarm vs Alarm on Threshold | 2 weeks CGM data with PA vs 2 weeks CGM data with AoT
  the difference in the percentage of time spent in 70-180 mg/dl range (TIR) between the Alarm on Threshold (AoT) and Predictive Alarm (PA) arms after 2 weeks of treatment (V2 vs V1 and V4 vs V3); the difference in the percentage of time spent above 250 mg/dl (TAR > 250 mg/dl) between the Alarm on Threshold and Predictive Alarm arms after 2 weeks of treatment (V2 vs V1 and V4 vs V3).
  the difference in main glucose metrics (%TIR, %TBR, %TAR) and glucose variability measures (SD, %CV, MAG, MAGE, HBGI, LBGI, ADRR, CONGA, MODD) between Group A (PA/AoT) and Group B (AoT/PA) at the end of the treatment period (V4) vs baseline (V1)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Diabetes and Metabolic Disorders Unit, Surgery, Dentistry, Paediatrics and Gynaecology, University of Verona, 1 Piazzale Stefani, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodbard D. Continuous Glucose Monitoring: A Review of Recent Studies Demonstrating Improved Glycemic Outcomes. Diabetes Technol Ther. 2017 Jun;19(S3):S25-S37. doi: 10.1089/dia.2017.0035. PMID 28585879
- [Background] Taleb N, Emami A, Suppere C, Messier V, Legault L, Chiasson JL, Rabasa-Lhoret R, Haidar A. Comparison of Two Continuous Glucose Monitoring Systems, Dexcom G4 Platinum and Medtronic Paradigm Veo Enlite System, at Rest and During Exercise. Diabetes Technol Ther. 2016 Sep;18(9):561-7. doi: 10.1089/dia.2015.0394. Epub 2016 Jun 29. PMID 27356172
- [Background] Christiansen MP, Garg SK, Brazg R, Bode BW, Bailey TS, Slover RH, Sullivan A, Huang S, Shin J, Lee SW, Kaufman FR. Accuracy of a Fourth-Generation Subcutaneous Continuous Glucose Sensor. Diabetes Technol Ther. 2017 Aug;19(8):446-456. doi: 10.1089/dia.2017.0087. Epub 2017 Jul 12. PMID 28700272
- [Background] Slover RH, Tryggestad JB, DiMeglio LA, Fox LA, Bode BW, Bailey TS, Brazg R, Christiansen MP, Sherr JL, Tsalikian E, Kaiserman KB, Sullivan A, Huang S, Shin J, Lee SW, Kaufman FR. Accuracy of a Fourth-Generation Continuous Glucose Monitoring System in Children and Adolescents with Type 1 Diabetes. Diabetes Technol Ther. 2018 Sep;20(9):576-584. doi: 10.1089/dia.2018.0109. Epub 2018 Jul 31. PMID 30063162
- [Background] Sherr JL, Tauschmann M, Battelino T, de Bock M, Forlenza G, Roman R, Hood KK, Maahs DM. ISPAD Clinical Practice Consensus Guidelines 2018: Diabetes technologies. Pediatr Diabetes. 2018 Oct;19 Suppl 27:302-325. doi: 10.1111/pedi.12731. No abstract available. PMID 30039513
- [Result] van Beers CA, DeVries JH, Kleijer SJ, Smits MM, Geelhoed-Duijvestijn PH, Kramer MH, Diamant M, Snoek FJ, Serne EH. Continuous glucose monitoring for patients with type 1 diabetes and impaired awareness of hypoglycaemia (IN CONTROL): a randomised, open-label, crossover trial. Lancet Diabetes Endocrinol. 2016 Nov;4(11):893-902. doi: 10.1016/S2213-8587(16)30193-0. Epub 2016 Sep 15. PMID 27641781
- [Result] Welsh JB, Gao P, Derdzinski M, Puhr S, Johnson TK, Walker TC, Graham C. Accuracy, Utilization, and Effectiveness Comparisons of Different Continuous Glucose Monitoring Systems. Diabetes Technol Ther. 2019 Mar;21(3):128-132. doi: 10.1089/dia.2018.0374. Epub 2019 Jan 25. PMID 30681379
- [Result] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583
- [Result] Wright LA, Hirsch IB. Metrics Beyond Hemoglobin A1C in Diabetes Management: Time in Range, Hypoglycemia, and Other Parameters. Diabetes Technol Ther. 2017 May;19(S2):S16-S26. doi: 10.1089/dia.2017.0029. PMID 28541136
- [Result] Stone MP, Agrawal P, Chen X, Liu M, Shin J, Cordero TL, Kaufman FR. Retrospective Analysis of 3-Month Real-World Glucose Data After the MiniMed 670G System Commercial Launch. Diabetes Technol Ther. 2018 Oct;20(10):689-692. doi: 10.1089/dia.2018.0202. Epub 2018 Aug 30. PMID 30160523
- [Result] Leelarathna L, Thabit H, Wilinska ME, Bally L, Mader JK, Pieber TR, Benesch C, Arnolds S, Johnson T, Heinemann L, Hermanns N, Evans ML, Hovorka R. Evaluating Glucose Control With a Novel Composite Continuous Glucose Monitoring Index. J Diabetes Sci Technol. 2020 Mar;14(2):277-283. doi: 10.1177/1932296819838525. Epub 2019 Mar 31. PMID 30931606
- [Derived] Marigliano M, Piona C, Mancioppi V, Morotti E, Morandi A, Maffeis C. Glucose sensor with predictive alarm for hypoglycaemia: Improved glycaemic control in adolescents with type 1 diabetes. Diabetes Obes Metab. 2024 Apr;26(4):1314-1320. doi: 10.1111/dom.15432. Epub 2024 Jan 4. PMID 38177091